CLINICAL TRIAL: NCT01340794
Title: A Phase 2 Study of Pazopanib (GW786034) in Patients With Advanced and Progressive Malignant Pheochromocytoma or Paraganglioma
Brief Title: Pazopanib Hydrochloride in Treating Patients With Advanced or Progressive Malignant Pheochromocytoma or Paraganglioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02588; NCI-2011-02588 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000699430; MAYO-MC107B; MC107B (Other: Mayo Clinic Cancer Center P2C); 8783 (Other: CTEP); N01CM00039 (NIH); N01CM00099 (NIH); N01CM62205 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Extra-Adrenal Paraganglioma; Metastatic Adrenal Gland Pheochromocytoma; Paraganglioma; Recurrent Adrenal Gland Pheochromocytoma
MeSH Terms: conditions — Paraganglioma, Extra-Adrenal; Pheochromocytoma; Paraganglioma | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pazopanib hydrochloride) (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-28 (days 1-14 of courses 1 and 2). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pazopanib Hydrochloride

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient

SUMMARY:
This phase II trial studies how well pazopanib hydrochloride works in treating patients with advanced or progressive malignant pheochromocytoma or paraganglioma. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the anti-tumor activity (in terms of the tumor response rate using the Response Evaluation Criteria in Solid Tumors [RECIST] criteria) of pazopanib (pazopanib hydrochloride) (GW786034) in patients with advanced malignant pheochromocytomas and paragangliomas.

SECONDARY OBJEC TIVES:

I. To assess safety profile of pazopanib. II. To assess duration of tumor response. III. To assess time to treatment failure. IV. To assess progression-free survival time. V. To assess overall survival time.

TERTIARY OBJECTIVES:

I. For patients with secretory tumors, to examine changes in urinary catecholamine and/or metanephrine levels.

II. For patients with secretory tumors, to examine whether pazopanib-induced changes in urinary catecholamine and/or metanephrine levels during the first cycle of treatment may be associated with objective tumor response.

III. To examine associations between tumor response and somatic mutational status in archived tumors, or germline mutational status in patient's peripheral blood mononuclear cells, (presence of succinate dehydrogenase complex subunit D [SDHD], succinate dehydrogenase complex subunit B [SDHB], ret proto-oncogene [RET], von Hippel-Lindau tumor suppressor [VHL], neurofibromatosis type-1).

IV. To examine associations between tumor response and tumor expression levels of angiogenic and vascular markers including hypoxia inducible factor 1, alpha (HIF-1a), vascular endothelial growth factor receptor (VEGF-R) (total and phospho-) and microvessel density in archival tumor tissue.

IV. To examine whether the extent of tumor response/regression may be correlated with plasma pazopanib (GW786034) concentration achieved after the third cycle (first cycle after run-in cycles) of pazopanib (GW786034) therapy.

OUTLINE:

Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-28 (days 1-14 of courses 1 and 2). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo urine and blood sample collection at baseline and periodically during study for correlative studies.

After completion of study therapy, patients are followed up every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant secretory or non-secretory pheochromocytoma or paraganglioma that is unresectable and deemed inappropriate for alternative local regional therapeutic approaches
* Objective evidence of tumor progression =< 185 days prior to registration as assessed by:

  * Unequivocal progression of objectively measured disease on successive appropriate imaging (e.g. computed tomography [CT] scan); in cases of uncertainty of tumor progression, the principal investigator of the study will be available to assist in decisions
* Measurable disease defined as:

  * At least one non-nodal lesion whose longest diameter can be accurately measured as >= 2.0 cm with chest x-ray, or as >= 1.0 cm with CT scan, CT component of a positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI); and/or
  * A lymph node whose short axis must be > 1.5 cm when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm)
  * Note: Tumor lesions in a previously irradiated area are not considered measurable disease
* Life expectancy > 24 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9 g/dL (5.6 mmol/L); transfusions not permitted =< 7 days of registration
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (except in cases of Gilbert's syndrome, where indirect bilirubin may be elevated, but the direct bilirubin remains within 1.5 x ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* NOTE: Subjects who have both bilirubin > ULN and AST/ALT > ULN are not eligible
* Alkaline phosphatase =< 2.5 x ULN
* Creatinine =< 1.5 mg/dL (133 umol/L) or within normal institutional limits OR creatinine clearance >= 50 mL/min/1.73m^2 for subjects with creatinine levels about institutional normal
* Urine protein/creatinine ratio =< 1 OR 24-hour urine < 1 gram
* Prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) =< 1.2 x ULN unless a subject is receiving Coumadin and has stable INR which is in range for the desired level of anticoagulation
* Blood pressure (BP) < 140 mmHg (systolic) and < 90 mmHg (diastolic); initiation or adjustment of BP medication is permitted prior to registration provided that the average of three BP readings at a visit prior to registration is < 140/90 mmHg

  * NOTE: All patients with secretory pheochromocytomas or paragangliomas are required to: 1) be evaluated in consultation by a hypertension specialist (at the registering institution) with experience in the management of hypertension in the setting of catecholamine-secreting tumors (usually an endocrinologist, nephrologist, or a cardiologist), and in the setting of hormone-associated hypertension 2) receive alpha- and beta-adrenergic blockade for at least 7 days prior to initiation of pazopanib (GW786034); the hypertension specialist of record for each patient should be committed to following the patient during the clinical study with evaluation by said specialist required at all run-in cycle evaluations (cycles 1 and 2) and also after the first continuous dosing cycle (cycle 3) and thereafter on an as needed basis
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to donate blood and tissue for correlative marker studies

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception NOTE: breastfeeding should be discontinued if the mother is treated with pazopanib (GW786034)
* Any of the following:

  * Chemotherapy/systemic therapy =< 4 weeks prior to registration
  * Radiotherapy =< 4 weeks prior to registration
  * Surgery =< 4 weeks prior to registration
  * Nitrosoureas or mitomycin C =< 6 weeks prior to registration
  * Those who have not recovered from adverse events due to agents administered more than 4 weeks earlier NOTE: Concurrent therapy with octreotide is allowed providing that tumor progression on this therapy has been demonstrated; concurrent therapy with bisphosphonates (e.g. zoledronic acid) or denosumab is also allowed.

NOTE: An unlimited number of prior chemotherapeutic or biologic therapies for malignant pheochromocytoma or paraganglioma is permitted; this includes prior anti-angiogenesis therapies such as tyrosine kinase inhibitors

* Any other ongoing investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib (GW786034) or other agents used in the study
* Any of the following:

  * Corrected QT (QTc) prolongation (defined as a QTc interval >= 500 msecs)
  * Left ventricular ejection fraction (LVEF) < institutional lower limit of normal (LLN)
  * Frequent ventricular ectopy
  * Evidence of ongoing myocardial ischemia
* Receiving prohibited cytochrome P450 (CYP) interactive concomitant medications within 7 days prior to registration
* Any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain pazopanib (GW786034)
* Receiving any medications or substances with risk of torsades de pointes; note: medications or substances with risk of torsades de pointes are prohibited; medications or substances with possible or conditional risk of torsades de pointes may be used while on study with extreme caution and careful monitoring; patients receiving these later cautionary agents must be monitored serially with electrocardiogram (ECG) weekly during the run-in and first cycle of therapy and at each evaluation thereafter NOTE: These medications should be discontinued or replaced with drugs that do not carry these risks, if possible
* Any of the following conditions:

  * Active peptic ulcer disease
  * Known intraluminal bowel metastatic lesions
  * Inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) or other gastrointestinal conditions which increase the risk of perforation
  * History of new abdominal fistula, gastrointestinal perforation or intra-abdominal abscess =< 84 days prior to registration; enrollment of patients with chronic/canalized fistulous tracts (present for > 84 days) is allowed
  * Serious or non-healing wound, ulcer, or bone fracture
  * History of familial QTc prolongation syndrome
* Any of the following conditions =< 185 days prior to registration:

  * Cerebrovascular accident (CVA) or transient ischemic attack (TIA)
  * Cardiac arrhythmia
  * Admission for unstable angina
  * Cardiac angioplasty or stenting
  * Coronary artery bypass graft surgery
  * Pulmonary embolism, untreated deep venous thrombosis (DVT) or DVT which has been treated with therapeutic anticoagulation < 42 days
  * Arterial thrombosis
  * Symptomatic peripheral vascular disease
  * Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
* Hemoptysis in excess of 2.5 mL (1/2 teaspoon) =< 60 days prior to registration
* Any of the following:

  * Known active and/or untreated brain metastases
  * Brain metastases requiring ongoing therapy (e.g. corticosteroids)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy
* Require heparin other than low-molecular weight heparin
* Prior use of pazopanib (GW786034)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Bible, Principal Investigator — Mayo Clinic Cancer Center P2C
Locations (11):
- United States (9):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota NCI Community Oncology Research Program, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Chinese University of Hong Kong-Prince of Wales Hospital, Shatin, Hong Kong
- National University Hospital Singapore, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened on 10/3/2011 and enrolled 2 patients prior to temporarily closing on 2/28/2012 due to safety concerns. After review of AEs, an addendum was implemented which instituted changes to treatment administration, namely, 2 - 14 day run-in periods where patients received pazopanib PO days 1-7 and then were assessed for safety.
Pre-assignment Details: A total of seven patients were recruited to this study. One of the 5 patients registered to the study post-addendum cancelled prior to initiating treatment.
Groups:
- Treatment: Pazopanib With no Run-in: Patients receive 800 mg pazopanib hydrochloride PO QD on days 1-28 of a 28 day cycle.
- Treatment: Pazopanib Run-in: Cycle 1:
  Patients receive 400 mg pazopanib hydrochloride PO QD on days 1-7 of a 14 day cycle.
  Cycle 2:
  Patients receive 800 mg pazopanib hydrochloride PO QD on days 1-7 of a 14 day cycle.
  Cycle 3 and beyond:
  Patients receive 800 mg pazopanib hydrochloride PO QD on days 1-28 of a 28 day cycle.
Period: Overall Study
Arm/Group | Treatment: Pazopanib With no Run-in | Treatment: Pazopanib Run-in
Started | 2 | 5
Completed | 2 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All 6 patients that began protocol treatment were included in the baseline analysis.
Groups:
- Treatment: Pazopanib Without Run-in: Patients receive 800 mg pazopanib hydrochloride PO QD on days 1-28 of a 28 day cycle.
- Treatment: Pazopanib With Run-in: Cycle 1:
  Patients receive 400 mg pazopanib hydrochloride PO QD on days 1-7 of a 14 day cycle.
  Cycle 2:
  Patients receive 800 mg pazopanib hydrochloride PO QD on days 1-7 of a 14 day cycle.
  Cycle 3 and beyond:
  Patients receive 800 mg pazopanib hydrochloride PO QD on days 1-28 of a 28 day cycle.
- Total: Total of all reporting groups
Arm/Group | Treatment: Pazopanib Without Run-in | Treatment: Pazopanib With Run-in | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Continuous [Median (Full Range); unit: years] | 42 [39 to 45] | 64.5 [53 to 80] | 57 [39 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR) (Complete Response [CR] or Partial Response [PR]) Using RECIST Version 1.1
Description: Response and progression are evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1) Ninety-five percent confidence intervals for the true response proportion was calculated using the exact binomial test.
  Complete Response (CR): All of the following must be true:
  1. Disappearance of all target and non-target lesions.
  2. Each lymph node must have reduction in short axis to <1.0 cm.
  Partial Response (PR):
  At least a 30% decrease in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking baseline measures as reference.
  Overall Response (OR) was calculated by summing the number of patients with a CR or PR.
Time Frame: Up to 5 years
Population: One of the two patients that initiated treatment with no run-in was found to be ineligible for this endpoint, leaving one patient evaluable for this endpoint in this treatment group. For patient confidentiality, results are not entered for endpoints based on 1 patient measures. All 4 patients that initiated treatment with a run-in were evaluable
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment: Pazopanib With no Run-in | Treatment: Pazopanib Run-in
Number analyzed (Participants) | 0 | 4
percentage of participants |  | 0 [0 to 60]

2. Secondary Outcome: Duration of Tumor Response
Description: Defined for all patients whose tumor met the criteria of CR or PR (using the RECIST criteria) as the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented.
Time Frame: Up to 5 years
Population: One of the two patients that initiated treatment with no run-in was found to be ineligible for this endpoint, leaving one patient evaluable for this endpoint in this treatment group. For patient confidentiality, results are not entered for endpoints based on 1 patient measures. None of the 4 patients that initiated treatment with a run-in responded
Arm/Group | Treatment: Pazopanib Without Run-in | Treatment: Pazopanib With Run-in
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival Time
Description: Overall survival time is defined as the time from registration to death due to any cause and will be estimated using the Kaplan-Meier method.
Time Frame: The time from registration to death due to any cause, assessed up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment: Pazopanib Without Run-in | Treatment: Pazopanib With Run-in
Number analyzed (Participants) | 0 | 4
months |  | 14.8 [7.6 to 26.3]

4. Secondary Outcome: Progression-free Survival Time
Description: Progression-free survival is defined as the time from registration to documentation of disease progression. If a patient dies without a documentation of disease progression, the patient will be considered to have had tumor progression at the time of their death unless there is sufficient documented evidence to conclude no progression occurred prior to death. Progression-free survival time will be estimated using the Kaplan-Meier method.
Time Frame: The time from registration to documentation of disease progression or death, whichever occurs first, assessed up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment: Pazopanib With no Run-in | Treatment: Pazopanib Run-in
Number analyzed (Participants) | 0 | 4
months |  | 6.5 [2.1 to 26.3]

5. Secondary Outcome: Time to Treatment Failure
Description: The time from the date of registration to the date at which the patient is removed from treatment due to progression, toxicity, or refusal, assessed up to 5 years.
Time Frame: Up to 5 years from registration
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment: Pazopanib With no Run-in | Treatment: Pazopanib Run-in
Number analyzed (Participants) | 0 | 4
months |  | 2.4 [0.8 to 5.7]

ADVERSE EVENTS:
Groups:
- Treatment: Pazopanib With Run-in: Patients receive 800 mg pazopanib hydrochloride PO QD on days 1-28 of a 28 day cycle.
Arm/Group | Treatment: Pazopanib Without Run-in | Treatment: Pazopanib With Run-in
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/4
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Pazopanib Without Run-in (N=2) | Treatment: Pazopanib With Run-in (N=4)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
CPK increased (Investigations) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
GGT increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Pazopanib Without Run-in (N=2) | Treatment: Pazopanib With Run-in (N=4)
Anemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (27) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (28) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (14) | 2 (7)
Vomiting (Gastrointestinal disorders) | 1 (12) | 1 (1)
Fatigue (General disorders) | 2 (32) | 4 (15)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (19) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (31) | 2 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1)
Hemoglobin increased (Investigations) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (17) | 0 (0)
Platelet count decreased (Investigations) | 2 (28) | 0 (0)
White blood cell decreased (Investigations) | 2 (25) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (7)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (6)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (33) | 1 (4)
Hypertension (Vascular disorders) | 2 (32) | 4 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less